CLINICAL TRIAL: NCT05735210
Title: Polso™ Watch BP Accuracy With BP Change Validation ChroniSense Study - IPPMed 1/2021
Brief Title: Polso™ Watch Blood Pressure Accuracy With Blood Pressure Change Validation
Acronym: BP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ChroniSense Medical Ltd. (Industry)
Collaborators: IPPMed, Institute for Pharmacology and Preventive Medicine GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Polso™ Watch BP Accuracy
Record Dates: First submitted 2023-01-29; First posted 2023-02-21 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Polso™ Watch blood pressure measurement compared to a reference blood pressure measurement (Experimental): Mean difference between the Polso™ Watch and reference measurement, and the associated standard deviation using data from the rest and induced change measurements following initialization
  Interventions: Device: Polso™ Watch blood pressure measurement compared to a reference blood pressure measurement

INTERVENTIONS:
Device: Polso™ Watch blood pressure measurement compared to a reference blood pressure measurement — The referenced blood pressure measurements are taken by dual auscultators.

SUMMARY:
Up to 185 adult test subjects to evaluate blood pressure measurement accuracy and stability of the Polso™ Watch compared to a reference blood pressure measurement.

DETAILED DESCRIPTION:
The purpose of this validation study is to assess, in an adult population, the three fundamental clinical tests:

1. Blood pressure measurement accuracy ("accuracy test")
2. Measurement accuracy after blood pressure change ("change test")
3. Blood pressure measurement accuracy throughout the specified stability-period ("stability test") To provide evidence that the device can track changes in blood pressure, this study includes study conditions that specifically induce changes in blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand and provide an informed consent to participate.
* Subject must be willing and able to comply with the study procedures.
* Subject must be ≥ 50 and <80 years of age.
* At least 30% of subjects shall be male and at least 30% of subjects shall be female.
* Subject with an arm circumference in the range of the reference device cuff selection.
* Subject with a wrist circumference in the range of the IMD wrist size selection.

Exclusion Criteria:

* Subjects with physical characteristics that (e.g. tattoos, scarification, unusual bone structure) may prevent proper application of the device under test.
* Subject is evaluated by the investigator or clinician and found to be medically unsuitable for participation in this study.
* Patients with known sustained or non-sustained ventricular/atrial arrhythmia (Ventricular tachycardia, supraventricular tachycardia, atrial fibrillation, bigeminy, and trigeminy), and left bundle branch block.
* Patients with implantable defibrillators, pacemakers, neurostimulators, or other implantable or worn devices which may interfere with the Polso™ Watch or be affected by the Polso™ Watch in normal operation and use.
* Patients with known Parkinson's disease, essential tremor, convulsive disorders, or other disorder which prevents them from keeping their forearm at rest.
* Patients with known elevated levels of Methemoglobin (MetHb) or Carboxyhemoglobin (COHb), or with anomalous hemoglobin.
* Patients with known severe anemia.
* Subjects with clinically apparent compromised circulation or peripheral vascular disease
* Subjects with clotting disorders or taking anticoagulants other than daily small doses of aspirin or similar
* Subjects that cannot tolerate sitting for up to 1 hour.
* Subjects that cannot perform the required blood pressure induced change procedure.
* Subject with a blood pressure (and other physiological parameters) demographic that has already been filled.
* Subjects with a known allergy to plastic, metals, and/or rubber.
* Subjects with a history of skin fragility or breakdown, such as ecchymosis or lacerations, affecting the upper extremities that would affect the application of non-invasive blood pressure cuff.
* Subjects who are pregnant.
* Subjects with BMI >35
* Subjects with BMI <20
* Subjects who gained or lost of >10% of their weight over a period of the last 6 months

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objectives: Main objective of the study is to evaluate blood pressure measurement accuracy and stability of the Polso™ Watch compared to a reference blood pressure measurement over time frame of 1 month average. | Through study completion, 1 month average
  Blood pressure measurements (units: mmHg) using the Polso™ Watch device will be taken and compared to reference blood pressure measurements taken at the same time using dual auscultatory blood pressure measurements, to show their accuracy and stability.

CONTACTS AND LOCATIONS:
Locations (1):
- IPPMed - Institute for Pharmacology and Preventive Medicine GmbH, Cloppenburg, Low Saxony, Germany

IPD SHARING:
Plan to Share IPD: No